CLINICAL TRIAL: NCT03777982
Title: A Randomized Phase III Study - Conventional Androgen Deprivation Therapy With or Without Abiraterone Acetate + Prednisone and Apalutamide Following a Detectable PSA After Radiation and Androgen Deprivation Therapy
Brief Title: Conventional Androgen Deprivation Therapy (ADT) With or Without Abiraterone Acetate + Prednisone and Apalutamide Following a Detectable PSA After Radiation and ADT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: PI is terminating the study due to slow/low accrual
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Principal Investigator, Anthony V. D'Amico, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-530
Record Dates: First submitted 2018-12-14; First posted 2018-12-19 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Prednisone; apalutamide; Abiraterone Acetate; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LHRH Agonist or Antagonist (Experimental): -LHRH agonist or antagonist should be prescribed per standard of care
  Interventions: Drug: LHRH Agonist or Antagonist
- Prednisone+Apalutamide+Abiraterone Acetate +LHRH Agonist (Experimental): * LHRH agonist or antagonist should be prescribed per standard of care
  * Abiraterone acetate will be taken once daily
  * Prednisone will be taken twice daily
  * Apalutamide will be taken once daily
  Interventions: Drug: Prednisone; Drug: Apalutamide; Drug: Abiraterone Acetate; Drug: LHRH Agonist or Antagonist

INTERVENTIONS:
Drug: Prednisone — Taking advantage of the anti-inflammatory properties of the medication, corticosteroids are used to decrease the swelling around tumors.
  Other Names: Deltasone
  Arms: Prednisone+Apalutamide+Abiraterone Acetate +LHRH Agonist
Drug: Apalutamide — Apalutamide also prevents the androgens from working within the prostate cancer cells, and can ultimately lead to cancer cell death.
  Other Names: ARN-509
  Arms: Prednisone+Apalutamide+Abiraterone Acetate +LHRH Agonist
Drug: Abiraterone Acetate — Abiraterone acetate interferes with an enzyme that is expressed in testicular, adrenal, and prostatic tumor tissues and is required as part of the body's androgen producing process. Because of this interference the amount of androgens produced are decreased. Abiraterone acetate, blocks androgen production at three sources; the testes, the adrenal glands, as well as from the tumor itself
  Other Names: Zytiga
  Arms: Prednisone+Apalutamide+Abiraterone Acetate +LHRH Agonist
Drug: LHRH Agonist or Antagonist — Luteinizing hormone-releasing hormone (LHRH) agonists (also called LHRH analogs or GnRH agonists) are drugs that lower the amount of testosterone made by the testicles
  Other Names: GnRH

SUMMARY:
This research study is being offered to those patients who have received radiation therapy and who are receiving long-term hormonal therapy for their prostate cancer and whose PSA remains detectable despite having received at least 6, but no more than 12 months of hormonal therapy.

The name of the study drugs involved in this study is:

* LHRHA (luteinizing hormone-releasing hormone agonist or antagonist)
* Abiraterone Acetate
* Apalutamide
* Prednisone

DETAILED DESCRIPTION:
This research study is a Phase III clinical trial. Phase III clinical trials test the effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that an intervention is being studied. In this study, the investigational agents are apalutamide and abiraterone acetate. Abiraterone acetate (used in combination with prednisone) is an FDA (the U.S. Food and Drug Administration) approved drug for prostate cancer, but is approved in patients that have prostate cancer spread to other parts of their body and have been previously treated with ADT. Apalutamide has also been approved by the FDA for men whose cancer does not respond to hormone therapy but it is still investigational for this type of cancer.

In this research study, the investigators are looking at two methods of androgen deprivation therapy (ADT), also known as hormonal therapy, to determine which method is better for improving long term cure rates. ADT blocks the function of hormones, including testosterone which prostate cancer uses to grow and spread. The first method of ADT includes prednisone, apalutamide, and abiraterone acetate plus standard ADT and the second method of ADT is standard ADT alone for men with this type of prostate cancer. Currently, the best standard treatment for men with this type of prostate cancer includes standard ADT. All participants in this study will receive the main standard form of ADT called a luteinizing hormone-releasing hormone agonist or antagonist (LHRHA).

ELIGIBILITY:
Inclusion Criteria:

* In order to ensure a homogenous population at study entry, a bone scan and not a PET will be used to ensure M0 high risk prostate cancer. A bone scan is to be done up to 6 months prior to the start of initial ADT therapy or up to one month after initiation of ADT to rule out bony metastatic disease.
* Histologically confirmed prostate cancer
* PSA> undetectable (any value at or above the lower limit of detection for the assay used) after radiation and at least 6, but not more than 12 months of conventional ADT (LHRH agonist or antagonist with or without oral anti androgens, excluding abiraterone acetate and apalutamide) in patients with non-metastatic high risk or N1 prostate cancer

  * High risk is defined per the NCCN guidelines - clinical, radiographic, or pathological (biopsy proven) T3 or higher, Gleason 8-10, PSA > 20 ng/mL, the presence of intraductal, ductal, or cribriform features with any Gleason score, and can be N0 or N1
  * A month is defined as 28 days
* Written informed consent and HIPAA authorization for release of personal health information prior to registration. NOTE: HIPAA authorization may be included in the informed consent or obtained separately. Subject must have the ability to understand and willingness to sign the written informed consent document.
* Age ≥18 at the time of consent
* ECOG Performance Status ≤ 2 (Appendix A)
* Demonstrate adequate organ function as defined in the table below. All screening labs to be obtained within 3 months of registration.
* System Laboratory Value
* Hematological:

  * Platelet count (plt)1 ≥ 100,000/ µL
  * Hemoglobin (Hgb)1 ≥ 9 g/dL
  * Absolute neutrophil count (ANC) ≥ 1000 cells/µL
* Renal:

  --CrCl2 ≥ 45 mL/min
* Hepatic and Other:

  * Bilirubin3 ≤ 1.5 × upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) < 2.5 × ULN
  * Alanine aminotransferase (ALT) < 2.5 × ULN
  * Serum Albumin > 3.0 g/dL
  * Serum potassium ≥ 3.5 mmol/L
* Coagulation:

  --International Normalized Ratio (INR) or Prothrombin Time (PT)
* Activated Partial Thromboplastin Time
* (aPTT) ≤ 1.5 × ULN (unless on prophylactic or therapeutic dosing with low molecular weight heparin)

  * Independent of transfusion and/or growth factors within 3 months prior to randomization
  * Cockcroft-Gault formula will be used to calculate creatinine clearance
  * In subjects with Gilbert's syndrome, if total bilirubin is >1.5 × ULN, measure direct and indirect bilirubin; if direct bilirubin is ≤1.5 × ULN, subject may be eligible
* Agrees to use a condom (even men with vasectomies) and another effective method of birth control if he is having sex with a woman of childbearing potential OR agrees to use a condom if he is having sex with a woman who is pregnant while on study drug and for 3 months following the last dose of study drug. Must also agree not to donate sperm during the study and for 3 months after receiving the last dose of study drug.
* Ability to understand and comply with study procedures for the entire length of the study as determined by the site investigator or protocol designee
* Medications known to lower the seizure threshold (section 5.4.4) must be discontinued or substituted prior to C1D1 of study treatment for patients on Arm 2
* Able to swallow pills

Exclusion Criteria:

* Prior radical prostatectomy (excluding TURP and simple prostatectomy)
* History of any of the following:

  * Seizure or known condition that may predispose to seizure (e.g., prior stroke within 1 year of randomization, brain arteriovenous malformation, Schwannoma, meningioma, or other benign CNS or meningeal disease which may require treatment with surgery or radiation therapy)
  * Severe or unstable angina, myocardial infarction, symptomatic congestive heart failure, arterial or venous thromboembolic events (eg, pulmonary embolism, cerebrovascular accident including transient ischemic attacks), or clinically significant ventricular arrhythmias within 6 months prior to randomization
* Known current evidence of any of the following:

  * Uncontrolled hypertension. Participants with a history of hypertension are allowed provided blood pressure is controlled by anti-hypertensive therapy
  * Gastrointestinal disorder affecting absorption
  * Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome.
  * Known active or chronic hepatitis B infection (defined as having a positive hepatitis B surface antigen (HBsAg) test at screening). Subject with past or resolved hepatitis B infection (defined as having a negative HBsAg test and positive antibody to hepatitis B core antigen test) are eligible. Hepatitis B viral DNA must be obtained in subjects with positive hepatitis B core antibody prior to first treatment start.
  * Active hepatitis C infection. Subjects positive hepatitis C antibody test are eligible if PCR is negative for hepatitis C viral DNA.
  * Pre-existing condition that warrants long-term corticosteroid use greater than the equivalent of 10 mg prednisone daily. Physiologic replacement is permitted. Topical, intra-articular steroids or inhaled corticosteroids are permitted.
  * Any condition that, in the opinion of the site investigator, would preclude participation in this study
  * Baseline moderate or severe hepatic impairment (ChildPugh Class B or C)
* Patients who are currently receiving treatment with a prohibited medication according to Section 5.4 (Tables 2 and 3), must discontinue that medication prior to starting treatment and must not restart for the duration of the study if randomized to ARM 2.
* Avoid co-administration of abiraterone acetate with CYP2D6 substrates that have a narrow therapeutic index. If an alternative treatment cannot be used, exercise caution and consider a dose reduction of the concomitant CYP2D6 substrate
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study drugs
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, psychiatric illness or social situations that would limit compliance with study requirements
* Individuals with a history of another malignancy are not eligible if the cancer is under active treatment or the cancer can be seen on radiology scans or if they are off cancer treatment but in the opinion of their oncologist have a high risk of relapse within 5 years.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2024-02-13 (Actual); Study Completion 2024-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony D'Amico, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (5):
- United States (5):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at Milford Regional Medical Center, Milford, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center in clinical affiliation with South Shore Hospital, South Weymouth, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor-Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication.
Access Criteria: Requests may be directed to: [contact information for Sponsor-Investigator or designee].

RESULTS

PARTICIPANT FLOW:
Groups:
- Prednisone+Apalutamide+Abiraterone Acetate +LHRH Agonist: * LHRH agonist or antagonist should be prescribed per standard of care
  * Abiraterone acetate will be taken once daily
  * Prednisone will be taken twice daily
  * Apalutamide will be taken once daily
  Prednisone: Taking advantage of the anti-inflammatory properties of the medication, corticosteroids are used to decrease the swelling around tumors.
  Apalutamide: Apalutamide also prevents the androgens from working within the prostate cancer cells, and can ultimately lead to cancer cell death.
  Abiraterone Acetate: Abiraterone acetate interferes with an enzyme that is expressed in testicular, adrenal, and prostatic tumor tissues and is required as part of the body's androgen producing process. Because of this interference the amount of androgens produced are decreased. Abiraterone acetate, blocks androgen production at three sources; the testes, the adrenal glands, as well as from the tumor itself
  LHRH Agonist or Antagonist: Luteinizing hormone-releasing hormone (LHRH) agonists (also called LHRH analogs or GnRH agonists) are drugs that lower the amount of testosterone made by the testicles
Period: Overall Study
Arm/Group | Prednisone+Apalutamide+Abiraterone Acetate +LHRH Agonist | LHRH Agonist or Antagonist
Started | 6 | 6
Completed | 6 | 5
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: Those who initiate the treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | LHRH Agonist or Antagonist | Prednisone+Apalutamide+Abiraterone Acetate +LHRH Agonist | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Median (Inter-Quartile Range); unit: years]
  Age | 70 [62 to 74] | 72 [66 to 74] | 71 [65 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 6 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 6 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
PSA pre-registration [Count of Participants; unit: Participants]
  PSA <0.5 ng/mL | 5 | 6 | 11
  PSA >=0.5 ng/mL | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Metastasis Free Survival
Description: the composite of metastasis or any cause death
Time Frame: 2 years
Population: The trial was terminated before the outcome measure data were collected.
Arm/Group | Prednisone+Apalutamide+Abiraterone Acetate +LHRH Agonist | LHRH Agonist or Antagonist
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: PSA Nadir
Description: PSA nadir is defined as the lowest PSA after RT completion
Time Frame: 2 years
Population: The trial was terminated before the outcome measure data were collected.
Arm/Group | Prednisone+Apalutamide+Abiraterone Acetate +LHRH Agonist | LHRH Agonist or Antagonist
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Castrate Resistant PSA Failure Free Survival
Description: Castrate resistant PSA failure is defined as the first PSA increase that is ≥ 25% and 2 ng/mL above the nadir, which is confirmed by a second value 3 or more weeks later, while the serum total testosterone level is < 50 ng/dl (per the PCWG2 criteria).
Time Frame: 2 years
Population: The trial was terminated before the outcome measure data were collected.
Arm/Group | Prednisone+Apalutamide+Abiraterone Acetate +LHRH Agonist | LHRH Agonist or Antagonist
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Prostate Cancer Specific Survival
Description: Prostate cancer specific survival is defined the time from randomization to death from prostate cancer where death due to other causes are considered as competing risk, or censored at the last date of follow up in living patients.
Time Frame: 2 years
Population: The trial was terminated before the outcome measure data were collected.
Arm/Group | Prednisone+Apalutamide+Abiraterone Acetate +LHRH Agonist | LHRH Agonist or Antagonist
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from randomization to death from any cause with men censored at time of last follow up if alive.
Time Frame: 2 years
Population: The trial was terminated before the outcome measure data were collected.
Arm/Group | Prednisone+Apalutamide+Abiraterone Acetate +LHRH Agonist | LHRH Agonist or Antagonist
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Disease Free Survival
Description: Disease free survival is measured from the date of randomization to the first recorded disease recurrence consisting of castrate resistant PSA failure and/or local, regional or distant failure and death from any cause, whichever comes first, or censored at the date of last disease assessment for those alive and disease recurrence free.
Time Frame: 2 years
Population: The trial was terminated before the outcome measure data were collected.
Arm/Group | Prednisone+Apalutamide+Abiraterone Acetate +LHRH Agonist | LHRH Agonist or Antagonist
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Toxicities were assessed every cycle. It was measured up to 3.8 years.
Description: Any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product, is medically important defined as a serious adverse event. All other events are defined as other adverse event.
Arm/Group | LHRH Agonist or Antagonist | Prednisone+Apalutamide+Abiraterone Acetate +LHRH Agonist
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LHRH Agonist or Antagonist (N=6) | Prednisone+Apalutamide+Abiraterone Acetate +LHRH Agonist (N=6)
Anemia (Blood and lymphatic system disorders) | 1 | 3
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 0 | 1
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Belching (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Fatigue (General disorders) | 3 | 6
Localized edema (General disorders) | 0 | 1
Pain (General disorders) | 1 | 1
Nail infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Creatinine increased (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 2
Platelet count decreased (Investigations) | 0 | 1
Weight gain (Investigations) | 1 | 1
White blood cell decreased (Investigations) | 0 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 2
Hyperlipidemia (Metabolism and nutrition disorders) | 0 | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 4
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Dizziness (Nervous system disorders) | 1 | 2
Dysgeusia (Nervous system disorders) | 0 | 1
Extrapyramidal disorder (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 2
Depression (Psychiatric disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 1
Libido decreased (Psychiatric disorders) | 1 | 1
Cystitis noninfective (Renal and urinary disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 1 | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 | 1
Renal calculi (Renal and urinary disorders) | 0 | 1
Urinary frequency (Renal and urinary disorders) | 2 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 1
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 | 1
Hot flashes (Vascular disorders) | 4 | 6
Hypertension (Vascular disorders) | 2 | 6
Hypotension (Vascular disorders) | 0 | 1
Vascular disorders - Other, specify (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-07): https://cdn.clinicaltrials.gov/large-docs/82/NCT03777982/Prot_SAP_000.pdf